CLINICAL TRIAL: NCT00380393
Title: A Study of the Efficacy Against Episodes of Clinical Malaria Due to P. Falciparum Infection of GSK Biologicals Candidate Vaccine RTS,S/AS01, Administered According to a 0,1,2-months Schedule in Children Aged 5 to 17 Months Living in Tanzania & Kenya
Brief Title: Efficacy of RTS,S/AS01 Vaccine Against Episodes of Malaria Due to P. Falciparum Infection in Children.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 106464
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2017-11

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium; RTS; S/AS01; Falciparum
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- GSK257049 Group (Experimental): Male or female subjects between 5 and 17 months of age at the time of first vaccination received 3 doses of GSK257049 vaccine administered intramuscularly in the left deltoid muscle at Days 0, 30 and 60.
  Interventions: Biological: GSK malaria vaccine 257049 Vaccine
- Rabipur Group (Active Comparator): Male or female subjects between 5 and 17 months of age at the time of first vaccination received 3 doses of Rabipur vaccine administered intramuscularly in the left deltoid muscle at Days 0, 30 and 60.
  Interventions: Biological: Sanofi-Pasteur's Human Diploid Cell Rabies Vaccine

INTERVENTIONS:
Biological: GSK malaria vaccine 257049 Vaccine — 3 dose intramuscular injection
  Other Names: RTS; S/AS01E vaccine
  Arms: GSK257049 Group
Biological: Sanofi-Pasteur's Human Diploid Cell Rabies Vaccine — 3 dose intramuscular injection
  Arms: Rabipur Group

SUMMARY:
This phase IIb trial is being done to find out if the RTS,S/AS01 vaccine helps to prevent children from falling ill with malaria and to evaluate vaccine safety.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child of between 5 months and 17 months of age at the time of first vaccination.
* Written or oral, signed or thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child..
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.

Exclusion Criteria:

* Acute disease at the time of enrolment.
* Serious acute or chronic illness determined by clinical or physical examination and laboratory screening tests.
* Laboratory screening tests for haemoglobin, total white cell count, platelets, ALT and creatinine out of acceptable limits.
* Planned administration/administration of a vaccine not foreseen by the study within 30 days of the first dose of vaccine(s) with the exception of tetanus toxoid or scheduled diphtheria, pertussis or measles vaccine.
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins, blood transfusions or other blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose
* Previous participation in any other malaria vaccine trial.
* Simultaneous participation in any other clinical trial.
* Same sex twin.
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 894 (Actual)
Dates: Start 2007-01-03 (Actual); Primary Completion 2008-08-15 (Actual); Study Completion 2008-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Kilifi, Kenya
- GSK Investigational Site, Amani, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bejon P, Lusingu J, Olotu A, Leach A, Lievens M, Vekemans J, Mshamu S, Lang T, Gould J, Dubois MC, Demoitie MA, Stallaert JF, Vansadia P, Carter T, Njuguna P, Awuondo KO, Malabeja A, Abdul O, Gesase S, Mturi N, Drakeley CJ, Savarese B, Villafana T, Ballou WR, Cohen J, Riley EM, Lemnge MM, Marsh K, von Seidlein L. Efficacy of RTS,S/AS01E vaccine against malaria in children 5 to 17 months of age. N Engl J Med. 2008 Dec 11;359(24):2521-32. doi: 10.1056/NEJMoa0807381. Epub 2008 Dec 8. PMID 19064627
- [Background] Lang TA, Gould J, von Seidlein L, Lusingu JP, Mshamu S, Ismael S, Liheluka E, Kamuya D, Mwachiro D, Olotu A, Njuguna P, Bejon P, Marsh V, Molyneux C. Approaching the community about screening children for a multicentre malaria vaccine trial. Int Health. 2012 Mar;4(1):47-54. doi: 10.1016/j.inhe.2011.10.003. PMID 24030880
- [Background] Lusingu J, Olotu A, Leach A, Lievens M, Vekemans J, Olivier A, Benns S, Olomi R, Msham S, Lang T, Gould J, Hallez K, Guerra Y, Njuguna P, Awuondo KO, Malabeja A, Abdul O, Gesase S, Dekker D, Malle L, Ismael S, Mturi N, Drakeley CJ, Savarese B, Villafana T, Ballou WR, Cohen J, Riley EM, Lemnge MM, Marsh K, Bejon P, von Seidlein L. Safety of the malaria vaccine candidate, RTS,S/AS01E in 5 to 17 month old Kenyan and Tanzanian Children. PLoS One. 2010 Nov 29;5(11):e14090. doi: 10.1371/journal.pone.0014090. PMID 21124768
- [Background] Olotu A, Lusingu J, Leach A, Lievens M, Vekemans J, Msham S, Lang T, Gould J, Dubois MC, Jongert E, Vansadia P, Carter T, Njuguna P, Awuondo KO, Malabeja A, Abdul O, Gesase S, Mturi N, Drakeley CJ, Savarese B, Villafana T, Lapierre D, Ballou WR, Cohen J, Lemnge MM, Peshu N, Marsh K, Riley EM, von Seidlein L, Bejon P. Efficacy of RTS,S/AS01E malaria vaccine and exploratory analysis on anti-circumsporozoite antibody titres and protection in children aged 5-17 months in Kenya and Tanzania: a randomised controlled trial. Lancet Infect Dis. 2011 Feb;11(2):102-9. doi: 10.1016/S1473-3099(10)70262-0. Epub 2011 Jan 13. PMID 21237715
- [Derived] Olotu A, Clement F, Jongert E, Vekemans J, Njuguna P, Ndungu FM, Marsh K, Leroux-Roels G, Bejon P. Avidity of anti-circumsporozoite antibodies following vaccination with RTS,S/AS01E in young children. PLoS One. 2014 Dec 15;9(12):e115126. doi: 10.1371/journal.pone.0115126. eCollection 2014. PMID 25506706
- [Derived] Warimwe GM, Fletcher HA, Olotu A, Agnandji ST, Hill AV, Marsh K, Bejon P. Peripheral blood monocyte-to-lymphocyte ratio at study enrollment predicts efficacy of the RTS,S malaria vaccine: analysis of pooled phase II clinical trial data. BMC Med. 2013 Aug 21;11:184. doi: 10.1186/1741-7015-11-184. PMID 23962071
- [Derived] Horowitz A, Hafalla JC, King E, Lusingu J, Dekker D, Leach A, Moris P, Cohen J, Vekemans J, Villafana T, Corran PH, Bejon P, Drakeley CJ, von Seidlein L, Riley EM. Antigen-specific IL-2 secretion correlates with NK cell responses after immunization of Tanzanian children with the RTS,S/AS01 malaria vaccine. J Immunol. 2012 May 15;188(10):5054-62. doi: 10.4049/jimmunol.1102710. Epub 2012 Apr 13. PMID 22504653
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Month 8 (Cross-sectional Visit)
Arm/Group | GSK257049 Group | Rabipur Group
Started | 447 | 447
Completed | 398 | 407
Not Completed | 49 | 40
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Migrated/moved from study area | 37 | 29
Not completed — Serious Adverse Event | 1 | 1
Not completed — Others | 5 | 4
Period: Month 14
Arm/Group | GSK257049 Group | Rabipur Group
Started | 447 | 447
Completed | 390 | 391
Not Completed | 57 | 56
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Migrated/moved from study area | 39 | 42
Not completed — Protocol Violation | 2 | 0
Not completed — Others | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK257049 Group | Rabipur Group | Total
Number analyzed (Participants) | 447 | 447 | 894
Age, Continuous [Mean (Standard Deviation); unit: Months] | 11.4 (3.6) | 11.4 (3.4) | 11.4 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 222 | 451
  Male | 218 | 225 | 443
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Frequency of First Case of Malaria Meeting the Primary Case Definition
Description: The first case of malaria meeting the primary case definition was defined as the first or only episodes with the presence of Plasmodium falciparum asexual parasitemia above (>) 2500 per microliter (μL) and the presence of fever greater than or equal to (≥) 37.5°C by active case detection (ACD) or passive case detection (PCD). Number of first case of malaria were assessed through estimate of vaccine efficacy (VE) adjusted or unadjusted for covariates, and are expressed in PYAR= number of episodes/Person Years at Risk.
Time Frame: Assessed over average of 7.8 months post Dose 3 (range 4.3 to 10.3 months)
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for efficacy, which included all evaluable for whom data concerning efficacy outcome measures were available.
Measure: Number; unit: PYAR
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 415 | 420
PYAR
  With estimate of VE adjusted for covariates: number analyzed (Participants) | 402 | 407
  With estimate of VE adjusted for covariates | 244.77 | 238.51
  With estimate of VE unadjusted for covariates | 249.23 | 242.06
Statistical Analysis 1: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p < 0.001, Regression, Cox; Vaccine Efficacy = 52.9, 95% CI 2-sided [28.1 to 69.1] — Point estimate of VE was adjusted for site, age, bednet use, area and distance from health center
Statistical Analysis 2: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p < 0.001, Regression, Cox; Vaccine Efficacy = 55.0, 95% CI 2-sided [31.4 to 70.4] — Point estimate of VE was not adjusted for site, age, bednet use, area or distance from health center

2. Secondary Outcome: Frequency of First Case Malaria Meeting the Secondary Case Definition
Description: The first case of malaria meeting the secondary case definition was defined as the first or only episodes with the presence of P.falciparum asexual parasitemia > 0 per μL and the presence of fever ≥ 37.5°C by active case detection (ACD) or passive case detection (PCD). Number of first case of malaria were assessed through estimate of vaccine efficacy (VE) adjusted or unadjusted for covariates, and are expressed in PYAR= number of episodes/Person Years at Risk.
Time Frame: Assessed over average of 7.8 months post Dose 3 (range 4.3 to 10.3 months)
Population: as for outcome 1
Measure: Number; unit: PYAR
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 415 | 420
PYAR
  With estimate of VE adjusted for covariates: number analyzed (Participants) | 402 | 407
  With estimate of VE adjusted for covariates | 244.72 | 237.21
  With estimate of VE unadjusted for covariates | 249.17 | 240.76
Statistical Analysis 1: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p < 0.001, Regression, Cox; Vaccine efficacy = 54.6, 95% CI 2-sided [31.2 to 70.0] — Point estimate of VE was adjusted for site, age, bednet use, area and distance from health center
Statistical Analysis 2: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p < 0.001, Regression, Cox; Vaccine efficacy = 56.5, 95% CI 2-sided [34.2 to 71.2] — Point estimate of VE was not adjusted for site, age, bednet use, area or distance from health center

3. Secondary Outcome: Multiple Events of Malaria Meeting the Primary Case Definition
Description: Multiple episodes of malaria meeting the primary case definition was defined as episodes with the presence of P.falciparum asexual parasitemia > 25000 per μL and the presence of fever ≥ 37.5°C by active case detection (ACD) or passive case detection (PCD). Number of primary case of malaria were assessed through estimate of vaccine efficacy (VE) adjusted or unadjusted for covariates, and are expressed in PYAR= number of episodes/Person Years at Risk.
Time Frame: Assessed over average of 7.8 months post Dose 3 (range 4.3 to 10.3 months)
Population: as for outcome 1
Measure: Number; unit: PYAR
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 415 | 420
PYAR
  With estimate of VE adjusted for covariates: number analyzed (Participants) | 402 | 407
  With estimate of VE adjusted for covariates | 253.69 | 255.36
  With estimate of VE unadjusted for covariates | 258.15 | 259.61
Statistical Analysis 1: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p = 0.0003, Regression, Cox; Vaccine efficacy = 55.8, 95% CI 2-sided [31.0 to 71.7] — Point estimate of VE was adjusted for site, age, bednet use, area and distance from health center
Statistical Analysis 2: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p < 0.001, Regression, Cox; Vaccine efficacy = 57.9, 95% CI 2-sided [34.3 to 73.0] — Point estimate of VE was not adjusted for site, age, bednet use, area and distance from health center

4. Secondary Outcome: Multiple Events of Malaria Meeting the Secondary Case Definition
Description: Multiple episodes of malaria meeting the secondary case definition was defined as episodes with the presence of P.falciparum asexual parasitemia > 0 per μL and the presence of fever ≥ 37.5°C by active case detection (ACD) or passive case detection (PCD). Number of secondary case of malaria were assessed through estimate of vaccine efficacy (VE) adjusted or unadjusted for covariates, and are expressed in PYAR= number of episodes/Person Years at Risk.
Time Frame: Assessed over average of 7.8 months post Dose 3 (range 4.3 to 10.3 months)
Population: as for outcome 1
Measure: Number; unit: PYAR
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 415 | 420
PYAR
  With estimate of VE adjusted for covariates: number analyzed (Participants) | 402 | 407
  With estimate of VE adjusted for covariates | 253.62 | 255.06
  With estimate of VE unadjusted for covariates | 258.07 | 259.31
Statistical Analysis 1: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p < 0.001, Regression, Cox; Vaccine efficacy = 58.0, 95% CI 2-sided [34.8 to 73.0] — Point estimate of VE was adjusted for site, age, bednet use, area and distance from health center
Statistical Analysis 2: Comparison: GSK257049 Group vs Rabipur Group; Vaccine efficacy against P. falciparum; Test type: Other; p < 0.001, Regression, Cox; Vaccine efficacy = 59.5, 95% CI 2-sided [37.1 to 73.9] — Point estimate of VE was not adjusted for site, age, bednet use, area and distance from health center

5. Secondary Outcome: Number of Subjects Positive for P. Falciparum Parasitaemia
Time Frame: At the Cross-Sectional Visit that took place for each participant at on average 7.8 months post Dose 3 (range 4.3 to 10.3 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 380 | 390
Participants | 7 | 11

6. Secondary Outcome: Geometric Mean Density of Asexual P. Falciparum Parasite
Description: Estimates of asexual P. falciparum parasite density were made at the investigator's sites according to laboratory standard operating procedures. Parasite density was presented as a geometric mean (GMean), expressed in parasite per microliters (μL).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: parasites/μL
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 380 | 390
parasites/μL | 1020 [135 to 7720] | 3486 [557 to 21813]

7. Secondary Outcome: Haemoglobin Values at Cross-Sectional Visit
Description: Haemoglobin values are expressed in grams per deciliter (g/dL).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 379 | 388
g/dL | 10.32 (1.01) | 10.37 (1.03)

8. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 swelling = swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants
  Any Pain, Dose 1 | 51 | 39
  Grade 3 Pain, Dose 1 | 0 | 0
  Swelling Pain, Dose 1 | 20 | 12
  Swelling 3 Pain, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 439 | 438
  Any Pain, Dose 2 | 45 | 38
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 439 | 438
  Grade 3 Pain, Dose 2 | 0 | 0
  Swelling Pain, Dose 2: number analyzed (Participants) | 439 | 438
  Swelling Pain, Dose 2 | 6 | 3
  Swelling 3 Pain, Dose 2: number analyzed (Participants) | 439 | 438
  Swelling 3 Pain, Dose 2 | 1 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 434 | 433
  Any Pain, Dose 3 | 76 | 80
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 434 | 433
  Grade 3 Pain, Dose 3 | 0 | 0
  Swelling Pain, Dose 3: number analyzed (Participants) | 434 | 433
  Swelling Pain, Dose 3 | 8 | 1
  Swelling 3 Pain, Dose 3: number analyzed (Participants) | 434 | 433
  Swelling 3 Pain, Dose 3 | 2 | 0
  Any Pain, Across doses | 143 | 130
  Grade 3 Pain, Across doses | 0 | 0
  Swelling Pain, Across doses | 30 | 13
  Swelling 3 Pain, Across doses | 3 | 0

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants
  Any Drowsiness, Dose 1 | 44 | 28
  Grade 3 Drowsiness, Dose 1 | 0 | 0
  Related Drowsiness, Dose 1 | 32 | 27
  Any Fever, Dose 1 | 55 | 138
  Grade 3 Fever, Dose 1 | 1 | 2
  Related Fever, Dose 1 | 49 | 133
  Any Irritability, Dose 1 | 26 | 12
  Grade 3 Irritability, Dose 1 | 0 | 0
  Related Irritability, Dose 1 | 17 | 8
  Any Loss of appetite, Dose 1 | 34 | 28
  Grade 3 Loss of appetite, Dose 1 | 0 | 1
  Related Loss of appetite, Dose 1 | 14 | 9
  Any Drowsiness, Dose 2: number analyzed (Participants) | 439 | 438
  Any Drowsiness, Dose 2 | 22 | 25
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 439 | 438
  Grade 3 Drowsiness, Dose 2 | 0 | 1
  Related Drowsiness, Dose 2: number analyzed (Participants) | 439 | 438
  Related Drowsiness, Dose 2 | 22 | 23
  Any Fever, Dose 2: number analyzed (Participants) | 439 | 438
  Any Fever, Dose 2 | 56 | 159
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 439 | 438
  Grade 3 Fever, Dose 2 | 3 | 8
  Related Fever, Dose 2: number analyzed (Participants) | 439 | 438
  Related Fever, Dose 2 | 51 | 156
  Any Irritability, Dose 2: number analyzed (Participants) | 439 | 438
  Any Irritability, Dose 2 | 16 | 7
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 439 | 438
  Grade 3 Irritability, Dose 2 | 0 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 439 | 438
  Related Irritability, Dose 2 | 14 | 7
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 439 | 438
  Any Loss of appetite, Dose 2 | 24 | 13
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 439 | 438
  Grade 3 Loss of appetite, Dose 2 | 0 | 1
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 439 | 438
  Related Loss of appetite, Dose 2 | 12 | 7
  Any Drowsiness, Dose 3: number analyzed (Participants) | 434 | 433
  Any Drowsiness, Dose 3 | 15 | 11
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 434 | 433
  Grade 3 Drowsiness, Dose 3 | 0 | 0
  Related Drowsiness, Dose 3: number analyzed (Participants) | 434 | 433
  Related Drowsiness, Dose 3 | 15 | 10
  Any Fever, Dose 3: number analyzed (Participants) | 434 | 433
  Any Fever, Dose 3 | 38 | 112
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 434 | 433
  Grade 3 Fever, Dose 3 | 1 | 2
  Related Fever, Dose 3: number analyzed (Participants) | 434 | 433
  Related Fever, Dose 3 | 32 | 107
  Any Irritability, Dose 3: number analyzed (Participants) | 434 | 433
  Any Irritability, Dose 3 | 17 | 2
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 434 | 433
  Grade 3 Irritability, Dose 3 | 0 | 0
  Related Irritability, Dose 3: number analyzed (Participants) | 434 | 433
  Related Irritability, Dose 3 | 13 | 1
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 434 | 433
  Any Loss of appetite, Dose 3 | 6 | 2
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 434 | 433
  Grade 3 Loss of appetite, Dose 3 | 0 | 0
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 434 | 433
  Related Loss of appetite, Dose 3 | 3 | 0
  Any Drowsiness, Across Doses | 66 | 59
  Grade 3 Drowsiness, Across Doses | 0 | 1
  Related Drowsiness, Across Doses | 55 | 56
  Any Fever, Across Doses | 125 | 268
  Grade 3 Fever, Across Doses | 5 | 12
  Related Fever, Across Doses | 111 | 262
  Any Irritability, Across Doses | 45 | 19
  Grade 3 Irritability, Across Doses | 0 | 0
  Related Irritability, Across Doses | 33 | 14
  Any Loss of appetite, Across Doses | 54 | 40
  Grade 3 Loss of appetite, Across Doses | 0 | 2
  Related Loss of appetite, Across Doses | 28 | 14

10. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 30-day (Days 0-29) post-vaccination follow-up period
Population: The analyses were performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants | 349 | 332

11. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the study period (Day 0 - Month 14)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants | 51 | 88

12. Secondary Outcome: Number of Subjects With Hemoglobin Values Outside Normal Ranges With Toxicity Grades
Description: Definitions for toxicity grading for hemoglobin were: Normal Hemoglobin = equal to or above (≥) 8.0 g/dL; Grade 1 Hemoglobin = under (<) 8.0 g/dL and above (>) 6.0 g/dL.; Grade 2 Hemoglobin = under (<) 6.0 g/dL.
Time Frame: At Day 0, Month 3 and at Cross-sectional Visit (took place between 7 and 13 months post Dose 1, mean: 10 months, standard deviation: 1.29)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants
  At Day 0: Normal | 445 | 446
  At Day 0: Grade 1 | 1 | 1
  At Day 0: Grade 2 | 1 | 0
  At Day 0: Missing | 0 | 0
  At Month 3: Normal | 410 | 413
  At Month 3: Grade 1 | 7 | 10
  At Month 3: Grade 2 | 0 | 0
  At Month 3: Missing | 30 | 24
  At Cross-sectional Visit: Normal | 391 | 397
  At Cross-sectional Visit: Grade 1 | 6 | 8
  At Cross-sectional Visit: Grade 2 | 0 | 0
  At Cross-sectional Visit: Missing | 50 | 42

13. Secondary Outcome: Number of Subjects With White Blood Cell (WBC) Values Outside Normal Ranges With Toxicity Grades
Description: Definitions for toxicity grading for WBC were: Normal WBC = ≥ 4.0 x 10^3 cells per microliters (cells/μL) or < 17 x 10^3 cells /μL; Grade 1 WBC = 2.5 to 4.0 x 10^3 cells/μL.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants
  At Day 0: Normal | 447 | 447
  At Day 0: Grade 1 | 0 | 0
  At Day 0: Missing | 0 | 0
  At Month 3: Normal | 416 | 422
  At Month 3: Grade 1 | 0 | 1
  At Month 3: Missing | 31 | 24
  At Cross-sectional Visit: Normal | 395 | 405
  At Cross-sectional Visit: Grade 1 | 0 | 0
  At Cross-sectional Visit: Missing | 52 | 42

14. Secondary Outcome: Number of Subjects With Platelet Values Outside Normal Ranges With Toxicity Grades
Description: Definitions for toxicity grading for platelets were: Normal Platelets = ≥ 75 x 10^3 cells/μL; Grade 1 Platelets = 50 to 74 x 10^3 /μL; Grade 2 Platelets = 25 to 49 x 10^3 /μL; Grade 3 Platelets = < 25 x 10^3 /μL.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants
  At Day 0: Normal | 445 | 447
  At Day 0: Grade 1 | 1 | 0
  At Day 0: Grade 2 | 0 | 0
  At Day 0: Grade 3 | 0 | 0
  At Day 0: Missing | 1 | 0
  At Month 3: Normal | 414 | 417
  At Month 3: Grade 1 | 1 | 0
  At Month 3: Grade 2 | 2 | 4
  At Month 3: Grade 3 | 0 | 1
  At Month 3: Missing | 30 | 25
  At Cross-sectional Visit: Normal | 386 | 396
  At Cross-sectional Visit: Grade 1 | 4 | 1
  At Cross-sectional Visit: Grade 2 | 1 | 0
  At Cross-sectional Visit: Grade 3 | 0 | 0
  At Cross-sectional Visit: Missing | 56 | 50

15. Secondary Outcome: Number of Subjects With Alanine Aminotransferase (ALT) Values Outside Normal Ranges With Toxicity Grades
Description: Definition for toxicity grading for ALT were: Normal ALT = ≤ 60 international units per liter (IU/L); Grade 1 ALT = 1.1 to 2.5 x Upper Limit of Normal (ULN); Grade 2 ALT = 2.6 to 5.0 x ULN.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants
  At Day 0: Normal | 446 | 447
  At Day 0: Grade 1 | 1 | 0
  At Day 0: Grade 2 | 0 | 0
  At Day 0: Missing | 0 | 0
  At Month 3: Normal | 413 | 420
  At Month 3: Grade 1 | 1 | 2
  At Month 3: Grade 2 | 0 | 1
  At Month 3: Missing | 33 | 24
  At Cross-sectional Visit: Normal | 393 | 397
  At Cross-sectional Visit: Grade 1 | 5 | 8
  At Cross-sectional Visit: Grade 2 | 0 | 1
  At Cross-sectional Visit: Missing | 49 | 41

16. Secondary Outcome: Number of Subjects With Creatinine Values Outside Normal Ranges With Toxicity Grades
Description: Definition for toxicity grading for creatinine were: Normal Creatinine = ≤ 60 micromols per liter (μmol/L); Grade 1 Creatinine = 1.1 to 1.5 x ULN; Grade 2 Creatinine = 1.6 to 3.0 x ULN.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 447 | 447
Participants
  At Day 0: Normal | 447 | 447
  At Day 0: Grade 1 | 0 | 0
  At Day 0: Grade 2 | 0 | 0
  At Day 0: Missing | 0 | 0
  At Month 3: Normal | 415 | 422
  At Month 3: Grade 1 | 0 | 0
  At Month 3: Grade 2 | 0 | 0
  At Month 3: Missing | 32 | 25
  At Cross-sectional Visit: Normal | 397 | 405
  At Cross-sectional Visit: Grade 1 | 1 | 0
  At Cross-sectional Visit: Grade 2 | 0 | 1
  At Cross-sectional Visit: Missing | 49 | 41

17. Secondary Outcome: Concentration of Antibodies Against the P. Falciparum Circumsporozoite (CS) Repeat Domain (Anti-CS)
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EU/mL).
Time Frame: as for outcome 12
Population: The analyses were performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 411 | 419
EU/mL
  At Day 0 | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.3]
  At Month 3: number analyzed (Participants) | 390 | 401
  At Month 3 | 539.6 [500.7 to 581.6] | 0.3 [0.3 to 0.3]
  At Cross-sectional Visit: number analyzed (Participants) | 366 | 384
  At Cross-sectional Visit | 71.9 [65.7 to 78.6] | 0.3 [0.2 to 0.3]

18. Secondary Outcome: Concentration of Antibodies Against Hepatitis B Surface Antigen (Anti-HBs)
Description: as for outcome 17
Time Frame: At Day 0 and at Month 3
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 410 | 419
EU/mL
  At Day 0 | 155.4 [134.6 to 179.5] | 187.4 [161.8 to 217.0]
  At Month 3: number analyzed (Participants) | 390 | 400
  At Month 3 | 46776.3 [39018.3 to 56076.8] | 168.0 [145.6 to 193.8]

19. Secondary Outcome: Frequency of Cluster of Differentiation 4 (CD4+) CS-specific T-cells
Description: T-cells expressing at least one of the following cytokines are presented here: interleukin-2 [IL-2], tumor-necrosis factor-alpha [TNF-α] and interferon-gamma [IFN-γ]. Frequency is expressed in cells/million, as assessed by Intracellular Cytokine Assay (ICA).
Time Frame: Prior to vaccination (Day 0)
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: cells/million
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 168 | 183
cells/million
  CD4-IFN-γ | 15 [1 to 55] | 14 [1 to 56]
  CD4-IL-2 | 111 [59 to 166] | 113 [53 to 212]
  CD4-TNF-α | 94 [40 to 218] | 92 [40 to 238]

20. Secondary Outcome: Frequency of Cluster of Differentiation 8 (CD8+) CS-specific T-cells
Description: as for outcome 19
Time Frame: Prior to vaccination (Day 0)
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: cells/million
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 161 | 165
cells/million
  CD8-IFN-γ | 1 [1 to 56] | 37 [1 to 90]
  CD8-IL-2 | 219 [117 to 417] | 222 [98 to 395]
  CD8-TNF-α | 100 [35 to 254] | 82 [37 to 203]

21. Secondary Outcome: Frequency of Cluster of Differentiation 4 (CD4+) CS-specific T-cells
Description: as for outcome 19
Time Frame: At Month 3
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: cells/million
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 156 | 169
cells/million
  CD4-IFN-γ | 33 [13 to 94] | 13 [1 to 79]
  CD4-IL-2 | 648 [359 to 1342] | 139 [66 to 463]
  CD4-TNF-α | 416 [225 to 755] | 172 [66 to 460]

22. Secondary Outcome: Frequency of Cluster of Differentiation 8 (CD8+) CS-specific T-cells
Description: as for outcome 19
Time Frame: At Month 3
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: cells/million
Arm/Group | GSK257049 Group | Rabipur Group
Number analyzed (Participants) | 143 | 156
cells/million
  CD8-IFN-γ | 36 [1 to 158] | 32 [1 to 160]
  CD8-IL-2 | 248 [131 to 428] | 219 [96 to 459]
  CD8-TNF-α | 201 [104 to 407] | 185 [68 to 390]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day post-vaccination period (Days 0-6), Unsolicited AEs: during the 30-day post-vaccination period(Days 0-29), SAEs: during the entire study period (Day 0 - Month 14).
Arm/Group | GSK257049 Group | Rabipur Group
All-Cause Mortality (participants affected / at risk) | 1/447 | 0/447
Serious Adverse Events (participants affected / at risk) | 51/447 | 88/447
Other Adverse Events (participants affected / at risk) | 385/447 | 396/447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049 Group (N=447) | Rabipur Group (N=447)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 11 (12)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cerebral malaria (Infections and infestations) | 0 (0) | 3 (3)
Cholera (Infections and infestations) | 1 (1) | 2 (2)
Dysentery (Infections and infestations) | 2 (2) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 10 (10) | 22 (22)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 8 (8) | 25 (25)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 16 (18) | 26 (28)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Schistosomiasis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 4 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Petroleum distillate poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Kwashiorkor (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Malignant mesenchymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 14 (17) | 20 (24)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049 Group (N=447) | Rabipur Group (N=447)
Decreased appetite (Metabolism and nutrition disorders) | 54 (64) | 40 (43)
Gastroenteritis (Infections and infestations) | 101 (120) | 81 (90)
Impetigo (Infections and infestations) | 27 (28) | 19 (20)
Irritability (Psychiatric disorders) | 45 (59) | 19 (21)
Lower respiratory tract infection (Infections and infestations) | 27 (27) | 28 (28)
Pain (General disorders) | 143 (172) | 130 (157)
Pneumonia (Infections and infestations) | 149 (195) | 141 (188)
Pyrexia (General disorders) | 125 (149) | 268 (409)
Rhinitis (Infections and infestations) | 27 (28) | 18 (20)
Somnolence (Nervous system disorders) | 66 (81) | 59 (64)
Swelling (General disorders) | 30 (34) | 14 (17)
Upper respiratory tract infection (Infections and infestations) | 81 (96) | 56 (59)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.